CLINICAL TRIAL: NCT04251273
Title: A Randomized Trial of a Text Message Quit Vaping Intervention for Young Adults
Brief Title: Text Message Quit Vaping Intervention for Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Truth Initiative (Other)
Responsible Party: Principal Investigator, Amanda L. Graham, PhD, Chief of Innovations, Truth Initiative
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TruthInitiativeQVS
Record Dates: First submitted 2020-01-23; First posted 2020-01-31 (Actual); Results first posted 2023-02-14 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-06

CONDITIONS: Tobacco Cessation
Keywords: E-cigarette Cessation; Vaping Cessation; Mobile Intervention; Digital Intervention
MeSH Terms: conditions — Tobacco Use Cessation

STUDY DESIGN:
Intervention Model Description: Arm 1: Intervention - Text message intervention Arm 2: Control - Assessment only
Who Masked: Participant
Masking Description: Participants are not explicitly told they are in the control group, although they may deduce their assignment from presence or lack of regular text message intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- This is Quitting (Experimental): Participants will be enrolled to receive messages from This is Quitting.
  Users receive one age-appropriate message per day tailored to their enrollment date or quit date, which can be set and reset via text message. Those not ready to quit receive 4 weeks of messages focused on building skills and confidence. Users who set a quit date receive messages for a week preceding it and 8 weeks afterward that include encouragement and support, skill- and self-efficacy building exercises, coping strategies, and information about the risks of vaping, benefits of quitting, and cutting down to quit. Keywords COPE, STRESS, SLIP, and MORE provide on-demand support.
  Interventions: Other: This is Quitting
- Assessment only Control (Other): After an initial enrollment message, participants will be contacted periodically to assess e-cigarette use. At the end of the intervention period, they will receive information on how to sign up for This is Quitting if they are interested in the program
  Interventions: Other: Assessment only Control

INTERVENTIONS:
Other: This is Quitting — Text message-based intervention for quit vaping support.
  Arms: This is Quitting
Other: Assessment only Control — Assessment only
  Arms: Assessment only Control

SUMMARY:
This research study, conducted by Truth Initiative, will help us learn how text messaging can help young adults between 18 and 24 years of age quit vaping.

DETAILED DESCRIPTION:
The Quit Vaping Study (QVS)'s primary aim is to conduct a fully powered comparative effectiveness trial to evaluate the effectiveness of a quit vaping text message program in promoting abstinence from e-cigarettes among young users aged 18-24. This study is a 2-arm randomized controlled trial conducted among young users aged 18-24 recruited through online channels. Participants will be randomized to a quit vaping text message intervention or to an assessment-only control condition and followed for 7 months to roughly correspond to 6-months post-treatment. The secondary aim is to examine potential mediators of program effectiveness, including treatment engagement and changes in self-efficacy and perceived social support for quitting.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-24
* Past 30-day use of e-cigarettes containing nicotine
* Interest in quitting e-cigarette use in the next 30 days
* US residence

Exclusion Criteria:

* Failure to confirm mobile number after initial sign-up

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2588 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2020-11-12 (Actual); Study Completion 2020-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda L Graham, PhD, Principal Investigator — Truth Initiative
Locations (1):
- Truth Initiative, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No
IPD are not available to other researchers. For access to deidentified dataset, please contact study administrator for more information.

REFERENCES:
- [Background] Graham AL, Jacobs MA, Amato MS, Cha S, Bottcher MM, Papandonatos GD. Effectiveness of a Quit Vaping Text Message Program in Promoting Abstinence Among Young Adult E-Cigarette Users: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2020 May 1;9(5):e18327. doi: 10.2196/18327. PMID 32356774
- [Background] Graham AL, Cha S, Papandonatos GD, Amato MS, Jacobs MA, Abroms LC, Berg CJ. E-cigarette and combusted tobacco abstinence among young adults: Secondary analyses from a U.S.-based randomized controlled trial of vaping cessation. Prev Med. 2022 Dec;165(Pt B):107119. doi: 10.1016/j.ypmed.2022.107119. Epub 2022 Jun 28. PMID 35777699
- [Result] Graham AL, Amato MS, Cha S, Jacobs MA, Bottcher MM, Papandonatos GD. Effectiveness of a Vaping Cessation Text Message Program Among Young Adult e-Cigarette Users: A Randomized Clinical Trial. JAMA Intern Med. 2021 Jul 1;181(7):923-930. doi: 10.1001/jamainternmed.2021.1793. PMID 33999133
- [Derived] Graham AL, Cha S, Do EK, Jacobs MA, Edwards G, Papandonatos GD. Dual abstinence from nicotine vaping and cannabis use among young people: secondary analyses from two U.S.-based randomized controlled trials of vaping cessation. Subst Abuse Treat Prev Policy. 2025 Nov 3;20(1):48. doi: 10.1186/s13011-025-00679-1. PMID 41177894

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment conducted from December 29, 2019 and March 18, 2020. Recruitment occurred online using advertisements on social media platforms.
Groups:
- This is Quitting: Participants will be enrolled to receive messages from This is Quitting.
  Users receive one age-appropriate message per day tailored to their enrollment date or quit date, which can be set and reset via text message. Those not ready to quit receive 4 weeks of messages focused on building skills and confidence. Users who set a quit date receive messages for a week preceding it and 8 weeks afterward that include encouragement and support, skill- and self-efficacy building exercises, coping strategies, and information about the risks of vaping, benefits of quitting, and cutting down to quit. Keywords COPE, STRESS, SLIP, and MORE provide on-demand support.
  This is Quitting: Text message-based intervention for quit vaping support.
Period: Overall Study
Arm/Group | This is Quitting | Assessment Only Control
Started | 1304 | 1284
Completed | 973 | 994
Not Completed | 331 | 290
Not completed — Lost to Follow-up | 331 | 290

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | This is Quitting | Assessment Only Control | Total
Number analyzed (Participants) | 1304 | 1284 | 2588
Age, Continuous [Mean (Standard Deviation); unit: Years] | 20.4 (1.7) | 20.4 (1.7) | 20.4 (1.7)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Female | 651 | 652 | 1303
  Gender: Male | 634 | 619 | 1253
  Gender: Non-binary or other | 18 | 8 | 26
  Gender: Unknown | 1 | 5 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 141 | 134 | 275
  Not Hispanic or Latino | 1163 | 1150 | 2313
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 11 | 7 | 18
  Asian | 71 | 52 | 123
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 19 | 38
  White | 1092 | 1067 | 2159
  More than one race | 72 | 90 | 162
  Unknown or Not Reported | 39 | 49 | 88
Region of Enrollment [Number; unit: participants]
  United States | 1304 | 1284 | 2588
Sexual orientation [Count of Participants; unit: Participants]
  Sexual minority | 243 | 250 | 493
  Not sexual minority (heterosexual) | 1061 | 1034 | 2095
Income [Count of Participants; unit: Participants]
  Live comfortably | 324 | 349 | 673
  Meet needs with a little left | 505 | 495 | 1000
  Just meet basic expenses | 399 | 379 | 778
  Don't meet basic expenses | 76 | 61 | 137
Student status [Count of Participants; unit: Participants]
  Current student | 976 | 956 | 1932
  Not current student | 328 | 328 | 656

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Self-reported 30-day Point Prevalence Abstinence (ITT)
Description: Number of participant who responded "No" to the question "In the past 30 days, did you vape at all, even a puff of someone else's?" Denominator is all randomized participants.
Time Frame: 7 months post enrollment
Population: All randomized participants (Intent-to-treat analysis)
Measure: Count of Participants; unit: Participants
Arm/Group | This is Quitting | Assessment Only Control
Number analyzed (Participants) | 1304 | 1284
Participants | 314 | 239

2. Secondary Outcome: Number of Participants With Self-reported 30-day Point Prevalence Abstinence (Responder Only)
Description: Number of participants with who responded 'No" to the question "In the past 30 days, did you vape at all, even a puff of someone else's?" Denominator is participants with responses only.
Time Frame: 7 month post enrollment
Population: 7 month assessment responders only (Responder Only)
Measure: Count of Participants; unit: Participants
Arm/Group | This is Quitting | Assessment Only Control
Number analyzed (Participants) | 976 | 995
Participants | 314 | 239

3. Secondary Outcome: Number of Participants With Self-reported 7-day Point Prevalence Abstinence (ITT)
Description: Number of participants who responded "No" to the question "Have you used any vape, even one puff, in the past 7 days?" Denominator is all randomized participants.
Time Frame: 7 months post enrollment
Population: All randomized participants (intent-to-treat analysis)
Measure: Count of Participants; unit: Participants
Arm/Group | This is Quitting | Assessment Only Control
Number analyzed (Participants) | 1304 | 1284
Participants | 440 | 385

4. Secondary Outcome: Number of Participants With Self-reported 7-day Point Prevalence Abstinence (Responder Only)
Description: Number of participants who responded "No" to the question "Have you used any vape, even one puff, in the past 7 days?" Denominator is those who responded to the question only.
Time Frame: 7 months post enrollment
Population: Only 7-month survey responders (responder only analysis)
Measure: Count of Participants; unit: Participants
Arm/Group | This is Quitting | Assessment Only Control
Number analyzed (Participants) | 973 | 994
Participants | 440 | 385

ADVERSE EVENTS:
Time Frame: Entire study duration (7-month participation)
Arm/Group | This is Quitting | Assessment Only Control
All-Cause Mortality (participants affected / at risk) | 0/1304 | 0/1284
Serious Adverse Events (participants affected / at risk) | 0/1304 | 0/1284
Other Adverse Events (participants affected / at risk) | 0/1304 | 0/1284

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-28): https://cdn.clinicaltrials.gov/large-docs/73/NCT04251273/Prot_SAP_000.pdf